CLINICAL TRIAL: NCT02560454
Title: Cognitive Training in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Acronym: TDAHEC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K140706
Record Dates: First submitted 2015-09-17; First posted 2015-09-25 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2018-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Cognitive Remediation; Working Memory Training; Cognitive training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cogmed® (Experimental): Cogmed® : working memory training (unifactorial) Before beginning the program an appointment of one hour will be organized to present the program.
  Participants will train at home during 25 sessions (about 30-45 minutes each) over a maximum of 5-6 weeks.
  A coach will call the participant one a week to verify program adherence. The coach will verify participant results on internet before calling.
  Interventions: Behavioral: Cogmed
- Presco® (Experimental): Presco® : different cognitive function are trained (multifactorial) Before beginning the program an appointment of one hour will be organized to present the program.
  Participants will train at home during 25 sessions (about 30-45 minutes each) over a maximum of 5-6 weeks.
  A coach will call the participant one a week to verify program adherence. The coach will verify participant results on internet before calling.
  Interventions: Behavioral: Presco
- Control (No Intervention): Control ( waiting list)

INTERVENTIONS:
Behavioral: Cogmed — Cogmed training working memory (unifactorial). Before beginning the program an appointment of one hour will be organized to present the program.
  Participants will train at home during 25 sessions (about 30-45 minutes each) over a maximum of 5-6 weeks.
  A coach will call the participant one a week to verify program adherence. The coach will verify participant results on internet before calling.
  Cogmed working memory training CogMed RM® (RoboMemo,Cognitive Medical Systems AB, Stockholm) version for children will be used in this program. Twelve exercises target verbal and visio-spatial working memory. Difficulty is adjusted depending on participant performance's
  Arms: Cogmed®
Behavioral: Presco — Presco drive of several cognitive functions (multifactorial). Before beginning the program an appointment of one hour will be organized to present the program.
  Participants will train at home during 25 sessions (about 30-45 minutes each) over a maximum of 5-6 weeks.
  A coach will call the participant one a week to verify program adherence. The coach will verify participant results on internet before calling.
  The program PRESCO® (Program in Cognitive Stimulation and rehabilitation ) comprises 40 exercises targeting: verbal and visio spatial working memory, attention capacities, reasoning, executive functioning , language and mental imagery. Only exercises targeting verbal, visual spatial working memory, and attentional capacities altered in ADHD are used in this present study. Difficulty is adjusted depending on the participant performances.
  Arms: Presco®

SUMMARY:
ADHD is associated with cognitive deficit. Therefore, cognitive training is often proposed as an intervention for ADHD that targets cognitive deficits, with specific exercises through intensive training sessions. This intervention is based on principles of brain plasticity and cerebral functional reorganizations.

Working memory deficits constitute a key impairment in ADHD. That is why, Cogmed working memory training is the most commonly used and studied cognitive training program in clinical practice and research. It is clear from most studies that Cogmed training program increases working memory in ADHD. However, transfer of learning is not demonstrated on: other cognitive functions that are not targeted by the program, on ADHD symptoms, nor on academic achievement.

In addition to this type of intervention multi-factorial program targeting different cognitive function as Presco also exist but have been less studied.

To address these challenges, this study will follow a randomized and controlled design.

The main objective of this study is to examine the impact of cognitive training in comparison with a control waiting-list group among children with ADHD on:

1. ADHD symptoms,
2. cognitive functioning,
3. attentional capacities
4. academic achievement.

The second objective is to compare two types of cognitive training a unifactorial program Cogmed targeting working memory and a multifactorial Presco focusing on different cognitive functions affected by ADHD.

Long-term effects are examined six months after training. Participants (n=90) will be randomly assigned to the two experimental group (Cogmed or Presco) or to the control group waiting list. Participants will be evaluated three time (time 1) just before the intervention, (time 2) six weeks after the first evaluation, immediately after the intervention and (time 3) six months after the intervention.

DETAILED DESCRIPTION:
Attention-Deficit Hyperactivity Disorder (ADHD) is a chronic developmental disorder characterized by symptoms of inattention, impulsivity and hyperactivity that do not correspond to the child's developmental level (American Psychiatric Association, 2013). For a diagnosis to be confirmed, symptoms must be present before age 12 and must be observed in at least to two domains of functioning, such as school, work, social interactions and family life (American Psychiatric Association, 2013).

ADHD is one of the most common neurobehavioral disorder with a prevalence estimated at about 5-7% for school-age children (Psychiatric Association, 2013).

ADHD alters family, social and academic functioning as well as one's professional life.

Results from studies indicated that working memory and inhibition are often altered in ADHD in childhood and persist into adulthood.

Pharmacological treatments of ADHD mostly include psychostimulants (Amphetamine and Methylphenidate) and non-stimulants (Atomoxetine, Clonidine, Guanfacine). Stimulants and no-stimulants are effective in managing ADHD symptoms.

However, these treatments present some limitation. For instance, comorbid disorders reduce stimulants efficacy in ADHD. Further, long-term effects over the year of stimulant are not yet known. Stimulants may cause side effects on sleep, hunger and growth. That is why some parents are reluctant to let their children take stimulants.

Currently, clinical guidelines recommend non-pharmacological interventions in conjunction with medication for the treatment of ADHD.

The above-mentioned limitations to the use of medication stress the importance of developing non-pharmacological approaches. Cognitive training is one type of non-pharmacological intervention used in ADHD.

This intervention consists in improving cognitive deficits through specific exercises during intensive training session. A growing number of studies examined the impact of cognitive training in ADHD.

Cognitive training is based on principles of brain plasticity with the aim to train cognitive function and to improve cognitive deficits in ADHD. According to these authors, during training changes occur in neural connection associated to ADHD. This modification allows far transfers to cognitive function not targeted by the program, to ADHD symptoms and academic performances.

Results from a meta-analysis indicated that 68% of 25 studies examining ADHD and cognitive training focus on working memory. These authors specify that Cogmed Working Memory Training is currently the most used and studied program. Indeed, this program is available in 25 countries and used by 150 clinical practitioners (http://www.cogmed.com).

Currently, one meta-analysis including seven studies examines Cogmed Working Memory Training program effects in ADHD. Results indicated that the impact of Cogmed on cognitive functioning, ADHD symptoms and academic performance remains controversial.

Cogmed is an unifactorial program targeting working memory. In addition to this type of intervention multi-factorial program targeting different cognitive function as Presco also exist but has been less studied.

Objectives To address these challenges, this study will follow a randomized and controlled design.

The main objective of this study is to examine the impact of cognitive training in comparison with a control group among children with ADHD on:

1. ADHD symptoms,
2. cognitive functioning,
3. attentional capacities
4. academic achievement.

The second objective is to compare two types of cognitive training a unifactorial program Cogmed targeting working memory and a multifactorial Presco focusing on different cognitive functions affected by ADHD.

Long-term effects are examined six months after training. Procedure Participants (n=90) will be randomly assigned to three groups.

1. Cogmed® : working memory training (unifactorial)
2. Presco® : different cognitive function are trained (multifactorial)
3. Control ( waiting list) Participants will be evaluated three time (time 1) just before the intervention, (time 2) six weeks after the first evaluation, immediately after the intervention and (time 3) six months after the intervention.

For Cogmed and Presco participants will train the same time. Before beginning the program an appointment of one hour will be organized to present the program.

Participants will train at home during 25 sessions (about 30-45 minutes each) over a maximum of 5-6 weeks.

A coach will call the participant one a week to verify program adherence. The coach will verify participant results on internet before calling.

Cogmed working memory training CogMed® (RoboMemo,Cognitive Medical Systems AB, Stockholm) version for children will be used in this program. Twelve exercises target verbal and visio-spatial working memory. Difficulty is adjusted depending on participant performance's The program PRESCO® (Program in Cognitive Stimulation and rehabilitation ) comprises 40 exercises targeting: verbal and visio spatial working memory, attention capacities, reasoning, executive functioning , language and mental imagery. Only exercises targeting verbal, visual spatial working memory, and attentional capacities altered in ADHD are used in this present study. Difficulty is adjusted depending on the participant performances.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 8 et ≤ 12, (2)
* ADHD diagnostic according to DSM IV or V criteria,
* score between 28 to 40 for The ADHD-RS,
* IQ-score, non-verbal reasoning (WISC-III or IV) ≥80, verbal reasoning (WISC-III or IV) ≥80,
* have internet and a computer at home,
* if methylphenidate treatments must not be changed for six months, (7) written consent by legal guardian.

Exclusion Criteria:

* Participant taking other medication than methylphenidate won't be included.
* Participant suffering from another neurological disorder than ADHD won't be included

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
The ADHD Rating Scale IV (ADHD RS) | 6 weeks

SECONDARY OUTCOMES:
ADHD Scale | 6 weeks and 6 months
  symptoms and psychopathology associated
TEA-Ch and Continuous Performance Test | 6 weeks and 6 months
  Attentional capacities
Behavior Rating Inventory of Executive Function (BRIEF) | 6 weeks and 6 months
  Cognitive functioning
Wechsler Test (WIAT-II CDN-F) | 6 weeks and 6 months
  Academic achievement

CONTACTS AND LOCATIONS:
Overall Officials: Amsellem Frédérique, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Amsellem, Paris, France